CLINICAL TRIAL: NCT01787058
Title: Monitoring and Evaluation Framework of the Dubai Cares' WASH in School Initiative
Brief Title: Evaluation of the Dubai Cares WASH in School Initiative
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: WaterAid (Other); Dubai Cares (Other); CARE (Unknown); Save the Children (Other); Oxfam (Unknown); UNICEF (Other)
Responsible Party: Principal Investigator, Matthew Freeman, MPH, PhD, Principal Investigator, Emory University
Other Study IDs: IRB00060756
Record Dates: First submitted 2013-02-01; First posted 2013-02-08 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Absenteeism; Diarrhea; Respiratory Tract Infections
Keywords: WASH; schoolchildren; absenteeism
MeSH Terms: conditions — Diarrhea; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dubai Cares beneficiary: Pupils who attend a school that has benefitted from a water, sanitation and hygiene intervention as part of the Dubai Cares program.
  Interventions: Other: Dubai Cares beneficiary
- Control: Pupils who attend a school of the same size and location as a school that benefitted from a water, sanitation and hygiene (WASH) intervention through the Dubai Cares program, but which has not benefitted from that program or any other WASH program since 2009.

INTERVENTIONS:
Other: Dubai Cares beneficiary — Installation or rehabilitation of school water points, latrines and hygiene kits; promotion of good WASH practices and behavior change at school and within the community; establishment of management systems to ensure sustained WASH financing, monitoring and maintenance.
  Groups: Dubai Cares beneficiary

SUMMARY:
This study will use longitudinal data collection to quantify the impact of a school-based water, sanitation and hygiene (WASH) program in Mali, West Africa, on pupil absenteeism, diarrheal illness, and respiratory illness.

Data will be collected from 100 intervention and 100 control schools across 4 regions in Mali. At each school research staff will randomly select 60 pupils in grades 3-6 (typically ages 7-14). Research staff will ask school directors to provide written consent for pupil participation in place of parents, a procedure that has been approved by the Malian Ministry of Education. Research staff will approach selected pupils at school to request informed oral assent for participation. The informed assent process and data collection will be conducted by local trained enumerators in the child's preferred language of French or Bambara. Oral rather than written assent was chosen due to varied literacy capabilities and to limit paperwork that identifies participants.

Data collection will take place at each school once every six to eight weeks during the duration of two school years. Research staff will conduct observations of school facilities, observations of handwashing behavior of children upon leaving latrines, and an interview with the school director about WASH conditions and school enrollment information. None of these school activities collect personal data or identifiers. Data collection with pupils will be done with the same pupils every 6-8 weeks and entails a 5-minute interview asking about recent absence and symptoms of diarrhea and respiratory illness.

All data collection will occur at the school, will be conducted by trained local enumerators, and will be stored on password-protected mobile data collection devices. Data will be uploaded to a password-protected server and will not contain personal identifying information. Enumerators will maintain a separate form that links pupil IDs with names, which will be kept confidential. There are no direct benefits other than contribution to general knowledge that will inform future school WASH projects. There are no risks to participation other than a small amount of class time missed by pupils, and great efforts will be made to minimize time outside of class.

DETAILED DESCRIPTION:
BACKGROUND AND SPECIFIC AIMS

Household-based water, sanitation and hygiene (WASH) improvements have demonstrated reductions in diarrheal. However, there is little academically sound research on the impact of school-based programs. The small body of current evidence is promising; school-based WASH interventions have been associated with reductions in absenteeism, particularly among girls. School WASH programs have also demonstrated decreases in diarrheal disease and helminth reinfection rates among school children.

In 2010, a consortium between UNICEF, CARE Mali, Oxfam GB, WaterAid Mali and Save the Children was launched to implement WASH programming in over 700 primary schools across Mali under the Dubai Cares WASH in Schools Initiative (DC Mali Initiative). Core activities of the project include: installing or rehabilitating school water points, latrines and hygiene kits; promoting good WASH practices and behavior change at school and within the community; and establishing management systems to ensure sustained financing, monitoring and maintenance.

The specific aim of this study is to quantify the impact of the DC Mali Initiative on pupil learning and health. Using longitudinal data collection, investigators will assess absenteeism, diarrhea, and respiratory infections in 100 intervention schools and compare the results to those observed in 100 control schools.

DATA COLLECTION ACTIVITIES

Facility Observations will be conducted by trained study enumerators using electronic data collection devices. The observations will be of the school facilities specifically, not of the students.

Structured Director Interviews will be administered to the school director. In the case where the school director is not available, an adjunct director with knowledge of school WASH facilities will be interviewed. Responses will be recorded on electronic data collection devices by trained enumerators. The questionnaire will address presence and functionality of school WASH facilities, and should take no more than 20 minutes. The information collected in this interview is a report on the state of facilities at the school and is not sensitive personal information.

Structured Pupil Interviews will be administered to a random sample of 40 pupils at each school. Pupils in grades 3-6 (typically ages 7-14) will be eligible for the sample. As this is a longitudinal study, the same pupils will be interviewed during each visit. New pupils will be selected at the start of the second academic year in September 2013 to replace those pupils who graduated or dropped out during the 2012-2013 academic year. Upon initial recruitment and after obtaining informed oral assent, pupil names will be recorded on a master list of participants, which will assign an ID to each participant. This list will be kept confidential by each enumerator. Enumerators will only record the corresponding ID number on data collection forms, and no names will be permanently recorded in the database. Pupil interview responses will be recorded on electronic data devices by trained enumerators. The interview will address recent history of school absenteeism, diarrheal illness, and respiratory illness. Pupils will also provide information about their age, grade, presence of a latrine at home, and academic grade the previous year. The pupil interview will take no more than five minutes per pupil. Interviews will be conducted in either French or the local language, according to the preference of the pupil.

A Roll Call will be taken of all pupils in the school on the day of each visit. Upon the first visit, enumerators will record a list of all pupils enrolled in the school. These lists with data will be kept confidential by enumerators and will not be shown to school administrators or others not involved in the research. At each data collection visit, enumerators will call the name of each pupil in the class and mark whether the pupil is absent. This method will be used to triangulate attendance data with school roster records. Aggregate data from all visits will be recorded in the database without any personal identifying information.

Handwashing observations will be made of pupils upon exiting latrines. Enumerators will observe the latrine area for 20 minutes and tally whether or not pupils use water and/or soap after leaving the latrine. No names or other personal or identifying information will be collected.

An Academic Data Review will be conducted three times throughout the 2012-13 and 2013-14 school years to determine percentage of children obtaining a passing average, percentage of children advancing to the next class, and percentage of drop-outs at each school. Only school-level data, disaggregated by gender and grade, will be collected during this review. No individual or personal data will be collected for this activity.

DATA MANAGEMENT AND MONITORING

This trial does not entail a medical intervention of any kind; therefore, a typical data safety and monitoring plan is not necessary. Study staff will be instructed to monitor any unforeseen situations that suggest an increase in risk to participants and immediately inform the study manager so that a decision can be made on how to mitigate those risks.

RISKS AND BENEFITS OF PARTICIPATION

Participation in the study will not subject participants to any excess risk other than a brief five-minute interruption of class time during classroom roll call, and a five-minute break from class for pupil participants to leave class for their interviews.

There are no direct benefits to participants other than knowing that information gained from this study will contribute to knowledge in the WASH sector worldwide about the educational and health impacts of improved WASH in schools. Schools participating as controls will be placed in high consideration by DC Mali Initiative partners for future interventions.

CONFIDENTIALITY

Names of pupil participants will be recorded separately from survey forms and will be destroyed after data collection has been completed. This information will only be retained on a separate ID linking form to ensure the same pupils are contacted in repeat visits to the school. Private health data relating recent history of diarrhea and respiratory illness will be linked to demographic information including age, gender, school, and school grade; however, this information will be insufficient to serve as an identifier. No identifiers will leave Mali

INFORMED CONSENT

The Malian Ministry of Education has granted a waiver of parental consent for pupil interviews. At each school, school directors will be asked to sign in loco parentis ("in the place of parent") on behalf of the pupil participants. These forms inform the director of the activities and purpose of the research and give permission to the researchers to carry out short interviews at the school with consenting pupils.

In addition to the loco parentis form, all pupil subjects selected to respond to the pupil interview will be read a full informed oral assent script the first time the interview is conducted. They will provide oral assent if they choose to participate in the longitudinal study. Continued assent will be obtained from pupils before commencing all subsequent data collection rounds. Oral assent rather than written has been chosen due to varying levels of literacy at the school as well as a desire to minimize paperwork that contains participants' names.

Investigators expect to sample 60 pupils per school. Therefore, school directors would sign the in loco parentis form for up to 60 pupils at each school. This form will be signed at the first visit, and will serve as consent for all subsequent visits. A total of 200 in loco parentis forms will be collected from school directors. A maximum of 12,000 oral assents will be recorded from the pupils during the first round of data collection, with an equal number of assents during each of the following data collection rounds.

ELIGIBILITY:
Inclusion Criteria:

* Attendance in a school that was randomly sampled from either the list of schools participating in the Dubai Cares water, sanitation and hygiene program or a list of non-program schools of the same size and in the same geographic area as a program school.
* In 3-6 grades

Exclusion Criteria:

* Inability to understand basic questions asked in French or one of three common local languages

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary school students attending public schools in the Koulikoro, Sikasso, Bamako, and Mopti regions of Mali
Sampling Method: Probability Sample
Enrollment: 10308 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Absenteeism rate | Every 6-8 weeks. Partcipants will be followed for 16 months (February 2013-June 2014)
  This indicator measures whether a pupil is absent on the day of a study staff visit. An all-school roll call will be used to measure single-day absenteeism for all pupils in grades 1-6. This indicator is collected longitudinally over the course of the trial with a time point every 6-8 weeks. Investigators will compare rates in intervention and control groups. This outcome is not a change outcome or a single outcome. It is a rate, which is a count of events over a specified period of time. This outcome measures more than one time point.

SECONDARY OUTCOMES:
7-day period prevalence of absenteeism | Every 6-8 weeks. Participants will be followed for 16 months (February 2013-June 2014)
  Schoolchildren will be asked to report the number of days they were absent from school in the past 7 days. This indicator is collected longitudinally over the course of the study every 6-8 weeks. Longitudinal prevalence ratios comparing intervention to control groups will be calculated.
7-day period prevalence of respiratory infection | Longitudinal prevalence: Baseline and every 6-8 weeks. Participants will be followed for 16 months (February 2013-June 2014)
  Schoolchildren from grades 3-6 will be asked whether they have experienced specific symptoms of respiratory infections in the last 7 days. This indicator is collected longitudinally over the course of the study every 6-8 weeks. Longitudinal prevalence ratios comparing intervention to control groups will be calculated.
2- and 7-day period prevalence of diarrhea | Longitudinal prevalence: Baseline and every 6-8 weeks. Participants will be followed for 16 months (February 2013-June 2014)
  Schoolchildren from grades 3-6 will be asked about the occurrence of diarrhea within the past 2 and 7 days. This indicator is collected longitudinally over the course of the study every 6-8 weeks. Longitudinal prevalence ratios comparing intervention to control groups will be calculated.
Prevalence of blood antibodies for enteric and neglected tropical diseases | Once, between February and March 2014
  School children between grades 1-6 will provide a capillary blood sample in the form of a dried blood spot (DBS). DBS will be shipped to a reference laboratory at the Centers for Disease Control and Prevention for analysis with a Luminex multiplexing assay. DBS will be analyzed for the presence of blood antibodies for a range of enteric and neglected tropical diseases, and results will be compared between intervention and control groups.

OTHER OUTCOMES:
Retention percentage | Baseline and every 6-8 weeks. Participants will be followed for 16 months (February 2013-June 2014)
  School attendance records and absenteeism roll call records (used for the primary study outcome) will be used to calculate the proportion of pupils who remain in school over the course of the study, comparing proportions in intervention and control groups.
Pass percentage | 3 months and 15 months (corresponding with end of school year June 2013 and June 2014)
  School records will be used to calculate the proportion of pupils who finish the school year with a passing exam score, comparing proportions in intervention and control groups.
Progression percentage | 3 months and 15 months (corresponding with end of school year June 2013 and June 2014)
  School attendance records and absenteeism roll call records will be used to calculate the proportion of pupils who progress to the next class between school years, comparing rates in intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Freeman, PhD, Principal Investigator — Emory University
Locations (1):
- Bamako, Sikasso, Koulikoro, and Mopti Regions, Bamako, Mali

REFERENCES:
- [Result] Trinies V, Garn JV, Chang HH, Freeman MC. The Impact of a School-Based Water, Sanitation, and Hygiene Program on Absenteeism, Diarrhea, and Respiratory Infection: A Matched-Control Trial in Mali. Am J Trop Med Hyg. 2016 Jun 1;94(6):1418-25. doi: 10.4269/ajtmh.15-0757. Epub 2016 Apr 25. PMID 27114292
- [Result] Chard AN, Trinies V, Moss DM, Chang HH, Doumbia S, Lammie PJ, Freeman MC. The impact of school water, sanitation, and hygiene improvements on infectious disease using serum antibody detection. PLoS Negl Trop Dis. 2018 Apr 16;12(4):e0006418. doi: 10.1371/journal.pntd.0006418. eCollection 2018 Apr. PMID 29659574
- [Derived] Rogier E, Moss DM, Chard AN, Trinies V, Doumbia S, Freeman MC, Lammie PJ. Evaluation of Immunoglobulin G Responses to Plasmodium falciparum and Plasmodium vivax in Malian School Children Using Multiplex Bead Assay. Am J Trop Med Hyg. 2017 Feb 8;96(2):312-318. doi: 10.4269/ajtmh.16-0476. Epub 2016 Nov 28. PMID 27895279